CLINICAL TRIAL: NCT06713031
Title: Prospective, Multicenter, Randomized Controlled Clinical Study of Medial Enhancement Technique for the Treatment of Old Femoral Neck Fractures
Brief Title: Medial Enhancement Technique for the Treatment of Old Femoral Neck Fractures
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Zhang Wei, Deputy head of orthopedics, Chinese PLA General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: S2024-342-01
Record Dates: First submitted 2024-11-16; First posted 2024-12-03 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-12

CONDITIONS: Fracture of Neck of Femur
Keywords: cannulated compression screws with iliac bone graft; Medial enhancement technique with iliac bone graft
MeSH Terms: conditions — Femoral Neck Fractures | interventions — Cycloserine

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cannulated compression screws + iliac bone graft group (Placebo Comparator)
  Interventions: Procedure: cannulated compression screws + iliac bone graft
- DCS + medial support plate + iliac bone graft group (Experimental)
  Interventions: Procedure: DCS + medial support plate + iliac bone graft

INTERVENTIONS:
Procedure: cannulated compression screws + iliac bone graft — Using "cannulated compression screws + iliac bone graft" technique to treat old femoral neck fractures
  Arms: Cannulated compression screws + iliac bone graft group
Procedure: DCS + medial support plate + iliac bone graft — Using "DCS + medial support plate + iliac bone graft" technique to treat old femoral neck fractures
  Arms: DCS + medial support plate + iliac bone graft group

SUMMARY:
A prospective, multi-center, randomized controlled study was conducted to validate the safety and effectiveness of employing the medial augmentation technique (incorporating the dynamic condylar screw and medial support plate) supplemented with bone grafting for the treatment of old femoral neck fractures.

ELIGIBILITY:
Inclusion Criteria:

1. Age >= 18 years, gender not specified;
2. Patients with femoral neck fractures who have not undergone surgery for more than 3 weeks, or patients with persistent non-union following internal fixation of femoral neck fractures;
3. Have indications for internal fixation surgery for femoral neck fractures and are able to tolerate the surgery;
4. Participants or their legal representatives are informed about the nature of this study and agree to participate.

Exclusion Criteria:

1. Participants who have not reached the primary endpoint of other drug, biological agent, or medical device clinical trials prior to enrollment;
2. Known history of hypersensitivity to one or more implanted materials by the patient;
3. Judged by the investigator as physically frail or unable to tolerate surgery due to other systemic diseases;
4. Active infectious foci in the hip joint or other parts of the body, as judged by the investigator;
5. Diagnosed with metabolic bone disease, radiation-induced bone disease, etc.;
6. Severe hip contracture deformity or severe muscle weakness that has been immobilized in functional position for a long time and painless;
7. Suffering from inflammatory arthritis, such as rheumatoid arthritis, systemic lupus erythematosus arthritis, ankylosing spondylitis, etc.;
8. Patients who lack the mental capacity or understanding to meet the requirements of participating in the study, or are difficult to cooperate with;
9. Other situations where the investigator deems the participant unsuitable for inclusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2024-12-10 (Estimated); Primary Completion 2024-12-10 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Fracture healing rate | 1 year

SECONDARY OUTCOMES:
Femoral head necrosis | 1 year
  Commonly used imaging tools include X-rays, Magnetic Resonance Imaging (MRI), and Computerized Tomography (CT). X-rays are the most commonly employed assessment tool, capable of displaying the morphology of the femoral head and whether the bone structure is normal. MRI and CT can provide more detailed images, aiding in the determination of the extent and range of femoral head necrosis.
Harris score | 1 year
  The Harris Score (Harris Hip Score, HHS) is a widely used scale for evaluating hip joint function and patient quality of life, often applied to assess the outcomes of hip replacement surgery or other treatments for hip joint diseases. It covers four main aspects: pain level, functional activity, joint range of motion, and hip joint deformity. The total score ranges from 0 to 100, with 100 being the best possible condition, indicating complete normalcy of hip joint function.
VAS score | 1 year
  The VAS score (Visual Analog Scale) is a commonly used tool for quantifying pain assessment that is suitable for measuring various degrees of pain. The VAS score typically employs a straight line 10 centimeters long (or an equivalent visual scale), with each end marked as "No Pain" and "Most Intense Pain" respectively. A straight line 10 centimeters long (or an equivalent visual scale) is often utilized, with each end labeled as "No Pain" and "Most Intense Pain."
Complications | 1 year
  Focusing on perioperative complications in patients, indications and symptoms of incision infection, including redness, swelling, drainage, and fever, should be carefully monitored. The incidence and severity of infection cases should be recorded and analyzed to evaluate the risk factors for postoperative infection and the effectiveness of preventive strategies. Unplanned reoperations should be recorded, including cases of primary surgery failure, development of complications, or other situations necessitating further surgical intervention. Detailed records of the causes, timing, and outcomes of reoperations will help evaluate the reliability of surgical techniques and internal fixation devices. Additionally, other postoperative complications, such as femoral head necrosis, repositioning of fracture ends, fixation loosening and breakage, should be meticulously recorded and observed.

CONTACTS AND LOCATIONS:
Locations (1):
- Chinese PLA General Hosptial, Beijing, China

IPD SHARING:
Plan to Share IPD: No